CLINICAL TRIAL: NCT02219594
Title: The Comparative Study of OCT，Gemstone CT and 320-detector Row Spiral CT for Evaluating Restenosis of Coronary Artery Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: W201310
Record Dates: First submitted 2014-08-10; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Heart Disease
Keywords: gemstone CT; 320-detector row spiral CT; optical coherence tomography(OCT); in-stent restenosis; coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemstone CT (Experimental): Gemstone CT ：Discovery CT750 HD（high definition） ，GE（General Electric Co.） Healthcare, Milwaukee； CT image for patient with suspected in-stent restenosis which Gemstone CT or 320-detector row spiral CT was assigned randomly to patient
  Interventions: Device: CT image for patient with suspected in-stent restenosis
- 320-detector row spiral CT (Active Comparator): 320-detector row spiral CT：Aquilion One, Toshiba, Nasu, Japan. CT image for patient with suspected in-stent restenosis which Gemstone CT or 320-detector row spiral CT was assigned randomly to patient .
  Interventions: Device: CT image for patient with suspected in-stent restenosis

INTERVENTIONS:
Device: CT image for patient with suspected in-stent restenosis — Gemstone CT or 320-detector row spiral CT was assigned randomly to patient who was suspected in-stent restenosis.About after 10 days,they would accept the check of OCT which wold be the "gold standard" of in-stent restenosis.
  Other Names: Gemstone CT; 320-detector row spiral CT; OCT

SUMMARY:
In-stent restenosis is a major reason of coronary heart disease recurrence .Even in drug eluting stent(DES), Restenosis rate could be up to 10% in diabetes and complex lesions though it was about 3-5% in general. It is particularly important that in-stent restenosis after implantation was early diagnosed and detected. The evaluation of OCT imaging is more accurate for narrow area calculation, more clear for narrow organization structure and more specific for detecting tissue types.It is currently the best way for restenosis histologic diagnosis.But it has many weakness such as the higher cost,an invasive test, expensive instrument, relatively complicated to operate,and etc.In this study, OCT image was regard as the "gold standard" of stent restenosis.

The improvement of spatial resolution of Gemstone CT can effectively improve the imaging quality and the measurement's accuracy of coronary artery stents.The diagnostic value of in-stent restenosis of Gemstone CT is higher than of the 320-detector row spiral CT. To a certain extent, the gemstone CT can replace OCT for examining the in-stent restenosis.

This study will examine the degree of in-stent restenosis by the gemstone CT and the 320-detector row spiral CT and compare the two ways on the basis of the result of OCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80， All genders
2. Unlimited time of implantation of coronary artery stents
3. Myocardial ischemia symptoms such as Chest tightness and/or chest pain in patients after stent implantation
4. No clinical symptoms, but myocardial ischemia suggested by other noninvasive tests
5. Routine re-testing 9-12 months after stent implantation.

Exclusion Criteria:

1. Renal insufficiency (serum creatinine > 120 umol/L)
2. Allergy of contrast
3. Severe heart failure
4. Uncontrollable heart rate or contraindication of taking metoprolol
5. Unstable condition
6. the ventricular rate beyond 70 beats / min and irregular rhythm after adjusting.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of detection of in-stent restenosis with the gemstone CT as compared to the 320-detector row spiral CT will be investigated | On the day in which a patient receives the gemstone CT and the 320-detector row spiral CT, estimated to take 10 mins
  Masked examiners (CT specialists) will evaluate and compare the degree of in-stent restenosis of the gemstone CT and the 320-detector row spiral CT images for the presence and features of in-stent restenosis. In this study, OCT image was regard as the "gold standard" of in-stent restenosis.

SECONDARY OUTCOMES:
Radiation burden of the the gemstone CT or the 320-detector row spiral CT and OCT | one month
  In a relatively short time,the patient will accept the two checks of CT and OCT(Interval period about 10 days).So,it is necessary to clear the reacts of these patients

OTHER OUTCOMES:
Measurement of the physical characteristics of in-stent restenosis structures seen on OCT | On the day in which a patient receives the check of OCT

CONTACTS AND LOCATIONS:
Overall Officials: Institute of Cardiovascular Disease Xuzhou Central Hospital, Study Director — Southeast University
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

REFERENCES:
- [Background] Colombo A, Latib A. [Treatment of drug-eluting stent restenosis with another drug-eluting stent: do not fail the second time!]. Rev Esp Cardiol. 2008 Nov;61(11):1120-2. No abstract available. Spanish. PMID 19000485
- [Background] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Background] Pasterkamp G, Falk E, Woutman H, Borst C. Techniques characterizing the coronary atherosclerotic plaque: influence on clinical decision making? J Am Coll Cardiol. 2000 Jul;36(1):13-21. doi: 10.1016/s0735-1097(00)00677-x. PMID 10898406
- [Background] Chau AH, Chan RC, Shishkov M, MacNeill B, Iftimia N, Tearney GJ, Kamm RD, Bouma BE, Kaazempur-Mofrad MR. Mechanical analysis of atherosclerotic plaques based on optical coherence tomography. Ann Biomed Eng. 2004 Nov;32(11):1494-503. doi: 10.1114/b:abme.0000049034.75368.4a. PMID 15636110
- [Background] Dewey M, Zimmermann E, Deissenrieder F, Laule M, Dubel HP, Schlattmann P, Knebel F, Rutsch W, Hamm B. Noninvasive coronary angiography by 320-row computed tomography with lower radiation exposure and maintained diagnostic accuracy: comparison of results with cardiac catheterization in a head-to-head pilot investigation. Circulation. 2009 Sep 8;120(10):867-75. doi: 10.1161/CIRCULATIONAHA.109.859280. Epub 2009 Aug 24. PMID 19704093
- [Result] Manfrini O, Slucca M, Bugiardini R. [Optical coherence tomography]. G Ital Cardiol (Rome). 2007 Jan;8(1):28-33. Italian. PMID 17354629
- [Result] Andreini D，Pontone G，Mushtaq S，et a1．Multidetector computed tomography coronary angiography for the assessment of coronary in-stent restenosis．Am J Cardiol，2010,105:645.